CLINICAL TRIAL: NCT02000089
Title: The Cancer of the Pancreas Screening-5 CAPS5)Study
Acronym: CAPS5
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH); American Association for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00087754; 1U01CA210170-01 (NIH); R01CA176828 (NIH)
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Pancreas Cancer; Peutz-Jeghers Syndrome (PJS); Gene Mutation; Germline Mutation Carrier; Lynch Syndrome
Keywords: familial pancreas cancer; (Peutz-Jeghers Syndrome) PJS; Breast cancer (BRCA) 2; Partner and Locator of BRCA2 (PALB2); Familial Atypical Multiple Mole- Melanoma (FAMMM); p16, CDKN2A; Breast Cancer (BRCA)1; (hereditary non-polyposis colorectal cancer or Lynch syndrome) HNPCC; Lynch Syndrome; hereditary pancreatitis; Protease Serine (PRSS); Chymotrypsin C (CTRC); Ataxia Telangiectasia Mutated(ATM)
MeSH Terms: conditions — Pancreatic Neoplasms; Peutz-Jeghers Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis; Breast Neoplasms; Dysplastic Nevus Syndrome; Hereditary pancreatitis; Hereditary Sensory and Autonomic Neuropathies | interventions — Secretin; CA-19-9 Antigen

STUDY DESIGN:
Intervention Model Description: Evaluation of the effect of diagnostic tests for pancreatic cancer
Masking Description: No masking of the diagnostic test results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Familial pancreas cancer relatives (Active Comparator): High Risk Group 2 (familial pancreatic cancer relatives):
  1. > 55 years old or 10 years younger than the age of youngest relative with pancreatic cancer, and
  2. come from a family with 2 or more members with a history of pancreatic cancer (2 of which have a first-degree relationship consistent with familial pancreatic cancer), and
  3. have a first-degree relationship with at least one of the relatives with pancreatic cancer.
  If there are 2 or more affected blood relatives, at least 1 must be a first-degree relative of the individual being screened
  Interventions: Drug: Secretin; Diagnostic Test: MRI; Other: Tumor marker gene test with CA19-9
- Group 1 germline mutation carrier (Active Comparator): High Risk Group 3 (Group 1 germline mutation carriers with an associated with an estimated lifetime risk of pancreatic cancer of ~10% or higher):
  a. > 50 years old or 10 years younger than the age of the youngest relative affected, if pancreatic cancer is in family, and b. The Patient is a carrier of a confirmed BRCA2, ATM or PALB2 mutation, regardless of family history of pancreatic cancer. b.> Individual is a carrier of a confirmed FAMMM (p16/CDKN2A) mutation, age 40 years or older, regardless of family history of pancreas cancer.
  Interventions: Drug: Secretin; Diagnostic Test: MRI; Other: Tumor marker gene test with CA19-9
- Group 2 germline mutation carrier (Active Comparator): High Risk Group 4 (Group 2 germline mutation carriers with an associated with an estimated lifetime risk of pancreatic cancer of ~5%):
  1. > 50 years old or 10 years younger than the age of the youngest relative with pancreatic cancer, and
  2. The patient is a carrier of a confirmed BRCA1 or HNPCC (hereditary non-polyposis colorectal cancer or Lynch syndrome, hMLH1, hMSH2, PMS1, hMSH6, EpCAM) gene mutation, and there is > 1 pancreatic cancer in the family, one of whom is a first- or second-degree relative of the subject to be screened.
  Interventions: Drug: Secretin; Diagnostic Test: MRI; Other: Tumor marker gene test with CA19-9
- Hereditary pancreatitis (Active Comparator): High risk group 5 (hereditary pancreatitis) with confirmed gene mutations that predispose to chronic pancreatitis, such as PRSS1, PRSS2, CTRC) and age 50 years or older (these patients have an estimated lifetime risk for pancreatic cancer of 40%) or twenty-years since their first attack of pancreatitis, whichever age is younger.
  Interventions: Drug: Secretin; Diagnostic Test: MRI; Other: Tumor marker gene test with CA19-9
- Peutz-Jeghers Syndrome (Active Comparator): 1. At least 30 years old, and
  2. at least 2 of 3 criteria diagnostic of Peutz-Jeghers syndrome (characteristic intestinal hamartomatous polyps, mucocutaneous melanin deposition, or family history of Peutz-Jeghers syndrome), or,
  3. known STK11 gene mutation carrier
  Interventions: Drug: Secretin; Diagnostic Test: MRI; Other: Tumor marker gene test with CA19-9
- Negative control (Active Comparator): 1. are undergoing routine EGD or Colonoscopy; or Endoscopic Ultrasound (EUS) and/or Endoscopic Retrograde Cholangiopancreatography (ERCP) for non-pancreatic indications as part of their standard medical care, and
  2. have no clinical or radiologic suspicion of pancreatic disease (chronic pancreatitis or pancreatic cancer)
  Interventions: Drug: Secretin
- Chronic Pancreatitis (Active Comparator): 1. are undergoing EUS and/or ERCP for evaluation and/or treatment of suspected or proven chronic pancreatitis as part of their standard medical care, and,
  2. have no clinical or radiologic suspicion of pancreatic cancer
  Interventions: Drug: Secretin
- Pancreas cancer (Active Comparator): a. are undergoing EUS and/or ERCP for evaluation and/or treatment of suspected or proven pancreatic ductal adenocarcinoma (based on clinical and radiologic evidence)
  Interventions: Drug: Secretin
- Pancreas cyst, IPMN evaluation (Active Comparator): are undergoing EUS and/or ERCP for evaluation and/or treatment of suspected or proven pancreatic cancer precursor, intraductal papillary mucinous neoplasm (based on clinical presentation and radiologic or prior EUS or radiologic evidence of a dilated main pancreatic duct and/or pancreatic cystic lesion communicating with the pancreatic ductal system).
  Interventions: Drug: Secretin

INTERVENTIONS:
Drug: Secretin — inject Secretin to stimulate pancreatic digestive fluid, which is collected in duodenum near ampulla via endoscope suction port. This fluid will be assessed for biomarkers.
  Other Names: ChiRhoStim
Diagnostic Test: MRI — MRI abdomen with contrast (MRCP) will be clinically indicated for abnormal novel CA-19-9 lab results.
  Other Names: MRCP
  Arms: Familial pancreas cancer relatives; Group 1 germline mutation carrier; Group 2 germline mutation carrier; Hereditary pancreatitis; Peutz-Jeghers Syndrome
Other: Tumor marker gene test with CA19-9 — A tumor marker gene test that will be used to stratify individuals into one of several circulating tumor marker reference ranges for CA19-9. The variants in the genes FUT3 and FUT2 affect the levels of CA19-9.
  Arms: Familial pancreas cancer relatives; Group 1 germline mutation carrier; Group 2 germline mutation carrier; Hereditary pancreatitis; Peutz-Jeghers Syndrome

SUMMARY:
Johns Hopkins clinical research office quality assurance group will monitor and audit this study at Johns Hopkins. The Sub Investigator at each site will be responsible for internal monitoring at their site.

DETAILED DESCRIPTION:
The Sub Investigator at each site will be responsible for internal monitoring at their site. The site sub Investigator and study team will report any serious adverse events to Principal Investigator and annually report adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Hereditary Pancreatitis or
* Peutz-Jeghers Syndrome or
* Strong family history of pancreas cancer on one side of the family tree or
* Confirmed germline mutation carrier (BRCA2, FAMMM (CDKN2A/p16), PALB2, BRCA1, ATM, HNPCC, Lynch Syndrome (hMLH1, hMSH2, PMS2, hMSH6, EpCAM) PRSS1, PRSS2, R122H, N291l, SPINK1, CFTR
* Endoscopic evaluation of pancreas scheduled

Exclusion Criteria:

* Medical comorbidities or coagulopathy that contraindicate endoscopy
* Prior surgery that prevent optimal endoscopic ultrasound such as partial or complete gastrectomy with Bilroth or Roux-en-Y anastomosis
* Stricture or obstruction in the upper GI tract that does not allow passage of the echoendoscope
* Poor performance status
* Inability to provide informed consent
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9000 (Estimated)
Dates: Start 2014-01-06 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate pancreatic juice for early cancer markers. | 10 years
  Aim #1: To evaluate pancreatic fluid mutations and circulating pancreatic epithelial cells as accurate markers of neoplasia by comparing their prevalence in cases with sporadic pancreatic neoplasia to healthy and disease controls.

SECONDARY OUTCOMES:
Compare pancreas juice with pancreas cyst fluid | 10 years
  Aim #2: To compare the prevalence of pancreatic fluid mutations and circulating pancreatic epithelial cells among a prospective cohort of individuals with sporadic pancreatic cysts undergoing pancreatic surveillance.

OTHER OUTCOMES:
Time disease progression and prevalence | 10 years
  Aim #3: To determine the prevalence of pancreatic lesions, pancreatic fluid mutations and circulating pancreatic epithelial cells among a large cohort of high-risk individuals undergoing pancreatic screening and surveillance of a new cohort in which screening is begun at age >55.
Diagnostic performance of a tumor marker gene test for CA19-9 interpretation | 5 years
  Aim #4 To evaluate the diagnostic performance of a tumor marker gene test to personalize the normal reference range of tumor markers such as CA19-9 for patients undergoing pancreatic surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goggins, MD, Principal Investigator — Johns Hopkins University
Locations (9):
- United States (9):
  - Yale University, New Haven, Connecticut
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Center, Harvard University, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Case Comprehensive Cancer Center, Case Western Medical Reserve, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumar S, Saumoy M, Oh A, Schneider Y, Brand RE, Chak A, Ginsberg GG, Kochman ML, Canto MI, Goggins MG, Hur C, Kastrinos F, Katona BW, Rustgi AK. Threshold Analysis of the Cost-effectiveness of Endoscopic Ultrasound in Patients at High Risk for Pancreatic Ductal Adenocarcinoma. Pancreas. 2021 Jul 1;50(6):807-814. doi: 10.1097/MPA.0000000000001835. PMID 34149034
- [Derived] Kohi S, Macgregor-Das A, Dbouk M, Yoshida T, Chuidian M, Abe T, Borges M, Lennon AM, Shin EJ, Canto MI, Goggins M. Alterations in the Duodenal Fluid Microbiome of Patients With Pancreatic Cancer. Clin Gastroenterol Hepatol. 2022 Feb;20(2):e196-e227. doi: 10.1016/j.cgh.2020.11.006. Epub 2020 Nov 5. PMID 33161160
- [Derived] Abe T, Koi C, Kohi S, Song KB, Tamura K, Macgregor-Das A, Kitaoka N, Chuidian M, Ford M, Dbouk M, Borges M, He J, Burkhart R, Wolfgang CL, Klein AP, Eshleman JR, Hruban RH, Canto MI, Goggins M. Gene Variants That Affect Levels of Circulating Tumor Markers Increase Identification of Patients With Pancreatic Cancer. Clin Gastroenterol Hepatol. 2020 May;18(5):1161-1169.e5. doi: 10.1016/j.cgh.2019.10.036. Epub 2019 Oct 30. PMID 31676359
- [Derived] Canto MI, Kerdsirichairat T, Yeo CJ, Hruban RH, Shin EJ, Almario JA, Blackford A, Ford M, Klein AP, Javed AA, Lennon AM, Zaheer A, Kamel IR, Fishman EK, Burkhart R, He J, Makary M, Weiss MJ, Schulick RD, Goggins MG, Wolfgang CL. Surgical Outcomes After Pancreatic Resection of Screening-Detected Lesions in Individuals at High Risk for Developing Pancreatic Cancer. J Gastrointest Surg. 2020 May;24(5):1101-1110. doi: 10.1007/s11605-019-04230-z. Epub 2019 Jun 13. PMID 31197699